CLINICAL TRIAL: NCT00956709
Title: Regional Anesthesia for Major Surgery of the Foot. Levobupivacaïne Ropivacaine 0.5% Versus 0.5% in the Sciatic Block Through médiofémorale
Acronym: SCIALERO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD/08/05-D
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Nerve Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levobupivacaïne 0,5 % (Active Comparator)
  Interventions: Drug: levobupivacaïne 0,5 %
- Ropivacaïne 0,5% (Active Comparator)
  Interventions: Drug: ropivacaïne 0,5 %

INTERVENTIONS:
Drug: levobupivacaïne 0,5 % — 20mL de levobupivacaïne 0,5 % 20mL de ropivacaïne 0,5 %
  Arms: Levobupivacaïne 0,5 %
Drug: ropivacaïne 0,5 % — 20mL de ropivacaïne 0,5 %
  Arms: Ropivacaïne 0,5%

SUMMARY:
Ropivacaine 0.5% and 0.5% in levobupivacaïne are used in regional anesthesia for major surgery of the foot. The literature does not highlight a significant difference in terms of onset of action between these two molecules to block the sciatic nerve [4]. Our hypothesis is that this lack of difference is due to the use of a neurostimulator for locating the injection site (indiscriminate nature of the anatomical approach to the sciatic nerve). Indeed, the sensitivity of neurostimulation is low compared with ultrasound [58] and ultrasound, for accurate visualization of the deposit of the local anesthetic around the nerve to improve the quality of the block and reduce the onset of action of local anesthetic [46, 47].

The investigators propose to make a comparative trial between levobupivacaïne 0.5% ropivacaine and 0.5% under the control of the ultrasound as part of a sciatic nerve block. The use of ultrasound will reduce the variability of results because the changes would be linked exclusively to the local anesthetic. The investigators test the hypothesis that levobupivacaïne gives better results in terms of onset of action than ropivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral major surgery of the foot: hallux valgus (not ambulatory), claw toes, fusion-Astragalo calcaneum, complex syntheses of tarsus-aged over 18 years .
* Male and female
* ASA 1 or 2
* Insured Social
* Informed Consent

Exclusion Criteria:

* Diabetes
* Intoxication-alcoholic chronic
* Allergy to local anesthetics
* Hemostasis disorders
* Hepatic failure
* Chronic pain syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levobupivacaïne 0,5 % | Ropivacaïne 0,5%
Started | 16 | 19
Completed | 16 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levobupivacaïne 0,5 % | Ropivacaïne 0,5% | Total
Number analyzed (Participants) | 16 | 19 | 35
Age, Continuous [Median (Full Range); unit: years] | 62 [36 to 83] | 62 [35 to 75] | 62 [35 to 83]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 15 | 25
  >=65 years | 6 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  France | 16 | 19 | 35

OUTCOME MEASURES:

1. Primary Outcome: Compare the Onset of Action of Ropivacaine 0.5% and levobupivacaïne 0.5 % for Sciatic Nerve Block Guided in Major Surgery of the Foot
Time Frame: 72 hours
Population: Two patients in each group had incomplete block before surgery.
Measure: Median (Full Range); unit: minutes
Arm/Group | Levobupivacaïne 0,5 % | Ropivacaïne 0,5%
Number analyzed (Participants) | 16 | 19
minutes | 40 [15 to 60] | 35 [10 to 60]
Statistical Analysis 1: Comparison: Levobupivacaïne 0,5 % vs Ropivacaïne 0,5%; Test type: Superiority or Other; p = 0.56, Wilcoxon (Mann-Whitney) — Two patients in each group had incomplete block before sugery

2. Secondary Outcome: Evaluate the Relative Position of the Tibial and Contigent Fibulaire Common in the Sciatic Nerve.
Time Frame: 72 hours
Reporting Status: Not Posted

3. Secondary Outcome: Duration of Motor Sciatic Block (h)
Time Frame: 72 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Levobupivacaïne 0,5 % | Ropivacaïne 0,5%
Number analyzed (Participants) | 16 | 19
hours | 15.54 [5.25 to 37.50] | 15.17 [4.42 to 20.50]
Statistical Analysis 1: Comparison: Levobupivacaïne 0,5 % vs Ropivacaïne 0,5%; Test type: Superiority or Other; p = 0.3354, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Duration of Sensory Sciatic Block (h)
Time Frame: 72 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Levobupivacaïne 0,5 % | Ropivacaïne 0,5%
Number analyzed (Participants) | 16 | 19
hours | 17.25 [6.25 to 53.50] | 15.00 [8.52 to 23.67]
Statistical Analysis 1: Comparison: Levobupivacaïne 0,5 % vs Ropivacaïne 0,5%; Test type: Superiority or Other; p = 0.0445, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Levobupivacaïne 0,5 % | Ropivacaïne 0,5%
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/19
Other Adverse Events (participants affected / at risk) | 0/16 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes